CLINICAL TRIAL: NCT02728908
Title: Detecting Traumatic Intracranial Hemorrhage With Microwave Technology - An Open Study Evaluating the Diagnostic Accuracy of a Microwave-based Device to Detect Traumatic Intracranial Hemorrhage (TICH), by Comparing Measurements on Trauma Patients With Confirmed vs Excluded TICH
Brief Title: Detecting Traumatic Intracranial Hemorrhage With Microwave Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hans Granhed (Other)
Collaborators: Medfield Diagnostics (Industry); Chalmers University of Technology (Other)
Responsible Party: Sponsor-Investigator, Hans Granhed, Sponsor-Investigator, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TICH 01
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Traumatic Intracranial Hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medfield Strokefinder MD100 — Measurement with Medfield Strokefinder MD100

SUMMARY:
An open study evaluating the diagnostic accuracy of a microwave-based device to detect traumatic intracranial hemorrhage (TICH), by comparing measurements on trauma patients with confirmed vs excluded TICH

DETAILED DESCRIPTION:
This open study will enrol trauma patients admitted to the Trauma Unit, Department of Surgery at Sahlgrenska University Hospital/Sahlgrenska. It will compare patients where TICH has been confirmed by CT (group A) to patients where CT has ruled out TICH (group B). Patients will be asked to participate in the study as early as possible after admission and CT scan. After physical examination, checking inclusion/exclusion criteria, and after informed consent has been acquired, the baseline microwave-based measurement will be performed. The diagnostic procedure is estimated to take 15 min; whereof total subject measurement time will be less than five minutes. Follow-up microwave measurements will be performed in conjunction with any follow-up CTs performed as part of the standard of care, during the hospitalized treatment period. If no follow-up CTs are performed as part of the standard of care, only the baseline microwave measurement will be performed.

Safety will be followed throughout the study, and a safety follow-up will be performed 12 hours after the last microwave-based investigation is finalized.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to Sahlgrenska University Hospital for trauma care.
* Patient deemed clinically stable.
* Patient should have a Glasgow Coma Scale rating of > 14
* TICH confirmed (group A) or ruled out (group B) by CT, performed within the latest 12 hours.
* Patient ≥ 18 years of age.
* Patient has signed the Informed Consent Form.

Exclusion Criteria:

* Patient has confirmed or suspected skull fracture.
* Patient has confirmed or suspected cervical spine fracture.
* The diagnostic procedure is deemed to interfere with the standard of care.
* Patient has a shunt or other foreign object implanted intracranially.
* Patient has agraffes/other metal parts, thick (> 1 cm) bandage, or other foreign materials attached to the head that are deemed to interfere with the diagnostic procedure.
* Any other condition or symptoms preventing the patient from entering the study, according to the Investigator's judgment.
* Females who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-04; Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
The diagnostic ability as measured by the area under receiver operating characteristic curve (AUC) of the device for detecting TICH | The diagnostic procedure has an estimated duration of 15 minutes
  The diagnostic ability of the device is calculated using a leave-one-out/n-fold cross-validation method

SECONDARY OUTCOMES:
The accuracy for estimating the position of the intracranial hemorrhage through a mathematical analysis of the microwave data | The diagnostic procedure has an estimated duration of 15 minutes
The accuracy for estimating the volume of the intracranial hemorrhage through a mathematical analysis of the microwave data | The diagnostic procedure has an estimated duration of 15 minutes
Mean time (± standard deviation) needed to complete the measurement procedure | The diagnostic procedure has an estimated duration of 15 minutes
Any adverse events occurring within 12 hours from the measurement procedure(s) | The diagnostic procedure has an estimated duration of 15 minutes, a safety follow-up will be performed 12 hours after the diagnostic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hans Granhed, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Department of Surgery, Trauma Unit
Locations (1):
- Sahlgrenska University Hospital, Department of Surgery, Trauma Unit, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No